CLINICAL TRIAL: NCT04269408
Title: A Phase IIb: Randomised, Single-Blind, Safety, Tolerability, Efficacy and Pharmacokinetic Study of NicaPlant® in Aneurysmal Subarachnoid Haemorrhage Patients Undergoing Aneurysm Clipping
Brief Title: A Safety and Efficacy Study of NicaPlant® in Aneurysmal Subarachnoid Haemorrhage Patients Undergoing Aneurysm Clipping
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BIT Pharma GmbH (Industry)
Collaborators: NeuroScios GmbH (Unknown); Data Magik Limited (Unknown); Pharm-Analyt Labor GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIT-002; 2017-005159-10 (EudraCT Number)
Record Dates: First submitted 2020-01-23; First posted 2020-02-13 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: NicaPlant; Nicardipine
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Nicardipine; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The clinical trial is defined as a single-blind study. For ethical reasons, no placebo implants will be used and therefore the surgeon cannot be blinded. All investigators/surgeons who have not been involved in the operation of a patient will remain blinded for this particular patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NicaPlant® (Experimental): 10 NicaPlant® implants (total 40 mg nicardipine) will be placed after clip ligation into the basal cisterns in direct contact with the exposed cerebral blood vessel walls.
  In addition patients will receive standard of care for aneurysmal subarachnoid haemorrhage patients according to the treatment guidelines.
  Interventions: Drug: Nicardipine; Other: Standard of care
- Control (Other): Standard of care for aneurysmal subarachnoid haemorrhage patients according to the treatment guidelines.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Nicardipine — 10 NicaPlant® implants releasing 4 mg nicardipine each.
  Other Names: NicaPlant®
  Arms: NicaPlant®
Other: Standard of care — Both arms receive the usual standard of care.

SUMMARY:
This study of NicaPlant® is conducted in patients who have a subarachnoid haemorrhage. Patients will be randomized in two treatment groups. Both groups will receive the standard of care and the investigational group will receive in addition NicaPlant®. NicaPlant® is tested to reduce the long-term complications of aneurysmal subarachnoid haemorrhage (aSAH).

DETAILED DESCRIPTION:
This is a safety, tolerability, efficacy and pharmacokinetic study of NicaPlant® in subarachnoid haemorrhage patients involving two treatment groups. Both treatment groups will receive standard of care and patients randomised to the investigational group will receive in addition NicaPlant® .

NicaPlant® is a nicardipine modified-release formulation. It is presented in the form of a rod-shaped implant with a 4 mg nicardipine load. Following aneurysm clip ligation, 10 NicaPlant® implants will be placed into the basal cisterns in direct contact with the exposed cerebral blood vessel walls.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained according to the Country regulation.
* Male or female patients aged 18 to 75 years (inclusive).
* World Federation of Neurological Surgeons (WFNS) grade III-IV.
* Ruptured saccular aneurysm, confirmed by angiography.
* Onset of aSAH clinical symptoms within the preceding 48 hours.
* Treatment of aneurysm via surgical clip ligation within 72 hours of aSAH is achievable.
* Female patients of child-bearing potential must have a negative pregnancy test (urine or serum) at screening and must agree to use adequate birth control up to 12 weeks after implantation of the study drug. Female patients are considered to be not of child-bearing potential if they have a history of tubal ligation or hysterectomy or are post-menopausal with a minimum of 2 years without a natural menstrual cycle. Male patients must agree to use adequate birth control up to 12 weeks after implantation of the study drug.

Exclusion Criteria:

* SAH due to other causes (e.g. trauma, fusiform or mycotic aneurysm).
* World Federation of Neurosurgery (WFNS) grade I, II and V patients.
* Pregnant or Lactating Women.
* Intraventricular or intracerebral blood, in the absence of subarachnoid blood.
* Treatment of aneurysm via endovascular embolisation.
* Presence of moderate or severe vasospasm on screening angiography.
* Any known or CT /MRI evidence of previous major cerebral damage
* Evidence of a cerebral infarction with neurological deficit on pre-treatment CT/MRI.
* History of malignant disease (except for non-melanoma skin cancer) within the previous 5 years or any history of malignant brain tumours or brain metastasis.
* Patients who have received an investigational product or participated in another interventional clinical study within 30 days prior to randomisation.
* Patients with known allergy for Poly(D,L-lactide-co-glycolide) (PLGA) or nicardipine.
* Major complication during aneurysm repair such as, but not limited to, massive intraoperative haemorrhage, brain swelling, or inability to secure the ruptured aneurysm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate to severe cerebral angiographic vasospasm assessed by digital subtraction angiography | day 8 ± 1 after aneurysm rupture
  Fishers Exact test
Safety by adverse event recording | trough study completion, an average of 2 years
  Descriptive summary

SECONDARY OUTCOMES:
Incidence of new cerebral infarcts on computer tomography (CT) of the brain versus post-intervention CT scan | up to day 14 ± 1 after aneurysm rupture
  Fishers exact test

OTHER OUTCOMES:
Incidence of vasospasm-related morbidity/mortality | within 21 days post aneurysm rupture
  Fishers exact test
Pharmacokinetic profile of NicaPlant® in plasma | within 21 days post aneurysm rupture or within hospitalisation if shorter
  AUC for multiple plasma samples
Nicardipine levels in cerebrospinal fluid (CSF) (only in patients provided with an external ventricular drain (EVD) at time of CSF removal for medical reasons) | within 21 days post aneurysm rupture or within hospitalisation if shorter
  Average concentration (Cav) for single CSF samples if sufficient CSF data is obtained.
Length of hospital stay | week 52 ± 2 after aneurysm rupture
  ANOVA
Modified Rankin Scale | week 12 ± 1 after aneurysm rupture
  Cochran-Mantel-Haenzel (CMH) test (with modified ridits)
  minimum value: 0, maximum value: 6, higher scores mean a worse outcome
Modified Rankin Scale | week 52 ± 2 after aneurysm rupture
  Cochran-Mantel-Haenzel (CMH) test (with modified ridits)
  minimum value: 0, maximum value: 6, higher scores mean a worse outcome
Glasgow Outcome Scale Extended | week 12 ± 1 after aneurysm rupture
  Cochran-Mantel-Haenzel (CMH) test (with modified ridits)
  minimum value: 1, maximum value: 8, higher scores mean a better outcome
Glasgow Outcome Scale Extended | week 52 ± 2 after aneurysm rupture
  Cochran-Mantel-Haenzel (CMH) test (with modified ridits)
  minimum value: 1, maximum value: 8, higher scores mean a better outcome
Montreal Cognitive Assessment | week 12 ± 1 after aneurysm rupture
  ANOVA
  minimum value: 0, maximum value: 30, higher scores mean a better outcome
Montreal Cognitive Assessment | week 52 ± 2 after aneurysm rupture
  ANOVA
  minimum value: 0, maximum value: 30, higher scores mean a better outcome
EQ-5D-5L | week 12 ± 1 after aneurysm rupture
  ANOVA
EQ-5D-5L | week 52 ± 2 after aneurysm rupture
  ANOVA
SF36 | week 12 ± 1 after aneurysm rupture
  ANOVA
SF36 | week 52 ± 2 after aneurysm rupture
  ANOVA

CONTACTS AND LOCATIONS:
Overall Officials: Claudius Thomé, Prof.Dr., Principal Investigator — Universitätsklinik Innsbruck, Universitätsklinik für Neurochirurgie
Locations (6):
- Austria (3):
  - Universitätsklinik Innsbruck, Universitätsklinik für Neurochirurgie, Innsbruck
  - Kepler Universitätsklinikum, Universitätsklinik für Neurochirurgie, Linz
  - Medizinische Universität Wien, Universitätsklinik für Neurochirurgie, Vienna
- Germany (3):
  - Charité Universitätsmedizin Berlin, Klinik für Neurochirurgie mit Arbeitsbereich pädiatrische Neurochirurgie, Berlin
  - Universitätsklinikum Göttingen, Neurochirurgische Klinik, Göttingen
  - Klinikum Rechts der Isar, Neurochirurgische Klinik und Poliklinik, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wessels L, Wolf S, Adage T, Breitenbach J, Thome C, Kerschbaumer J, Bendszus M, Gmeiner M, Gruber A, Mielke D, Rohde V, Wostrack M, Meyer B, Gempt J, Bavinzski G, Hirschmann D, Vajkoczy P, Hecht N. Localized Nicardipine Release Implants for Prevention of Vasospasm After Aneurysmal Subarachnoid Hemorrhage: A Randomized Clinical Trial. JAMA Neurol. 2024 Oct 1;81(10):1060-1065. doi: 10.1001/jamaneurol.2024.2564. PMID 39158893